CLINICAL TRIAL: NCT01249027
Title: XIENCE V Everolimus Eluting Coronary Stent System (EECSS) China: Post-Approval, Single-Arm Study
Acronym: XV CHINA SAS
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-388
Record Dates: First submitted 2010-11-24; First posted 2010-11-29 (Estimated); Results first posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2018-10

CONDITIONS: Angioplasty; Chronic Coronary Occlusion; Stent Thrombosis; Vascular Disease; Myocardial Ischemia; Coronary Artery Stenosis; Coronary Disease; Coronary Artery Disease; Coronary Restenosis
Keywords: Drug eluting stents; Stents; China; DES; XIENCE V EECSS
MeSH Terms: conditions — Vascular Diseases; Myocardial Ischemia; Coronary Stenosis; Coronary Disease; Coronary Artery Disease; Coronary Restenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: Single arm prospective, observational, single-arm, open-label, multicenter, postapproval registry study using XIENCE V® Everolimus Eluting Coronary Stent System (EECSS).
  Interventions: Device: XIENCE V® Everolimus Eluting Coronary Stent System (EECSS)

INTERVENTIONS:
Device: XIENCE V® Everolimus Eluting Coronary Stent System (EECSS) — Patients who receive XIENCE V® Everolimus Eluting Coronary Stent System (EECSS)will be invited to participate in the study.

SUMMARY:
This is a prospective, observational, single-arm, open-label, multicenter, postapproval registry study in China. The purpose of this study is to:

* Evaluate the continued safety and effectiveness of the XIENCE V EECSS in a cohort of real-world patients receiving the XIENCE V EECSS during commercial use
* Evaluate patient compliance to dual antiplatelet therapy (DAPT)

ELIGIBILITY:
Inclusion Criteria:

* The patient or patient's legally-authorized representative agrees to participate in this study by signing the Ethics Committee-approved informed consent form (ICF).
* Only XIENCE V stent(s) is/are implanted into the coronary vasculature during the index procedure.

Exclusion Criteria:

* The inability to obtain a signed ICF

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: General Chinese interventional cardiology population
Sampling Method: Non-Probability Sample
Enrollment: 2605 (Actual)
Dates: Start 2010-11; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, MB, MSc, MD, FACC, FESC, FSCAI, Principal Investigator — Fudan University; Jiyan Chen, MD, Principal Investigator — Institute of Cardiovascular Guangdong, Guangdong Provincial People's Hospital; YuJie Zhou, MD, Ph.D, Principal Investigator — An Zhen Hospital
Locations (1):
- Abbott Vascular, Santa Clara, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: XIENCE V China SAS was designed to enroll approximately 2500 patients. The first patient was enrolled on November 26, 2010. The enrollment was completed on December 10, 2011, with a total of 2605 patients enrolled at 53 sites. Of 2605 patients, a total of 123 subjects were withdrawn. Per protocol population is 2482.
Pre-assignment Details: A total of 123 subjects were withdrawn due to following reasons: 82 subjects had incomplete informed consent procedures;11 subjects enrolled repeatedly;1 subject did not have a stent at the starting point for surgery;18 subjects surgically implanted with other stents at the start;1 subject withdrew informed consent;10 subjects deregistered.
Period: 1 Year Clinical Follow up
Arm/Group | Observational
Started | 2482
Completed | 2391
Not Completed | 91
Period: 2 Years Clinical Follow up
Arm/Group | Observational
Started | 2391
Completed | 2254
Not Completed | 137
Period: 3 Years Clinical Follow up
Arm/Group | Observational
Started | 2254
Completed | 2223
Not Completed | 31
Period: 4 Years Clinical Follow up
Arm/Group | Observational
Started | 2223
Completed | 2210
Not Completed | 13
Period: 5 Years Clinical Follow up
Arm/Group | Observational
Started | 2210
Completed | 2142
Not Completed | 68

BASELINE CHARACTERISTICS:
Arm/Group | Observational
Number analyzed (Participants) | 2482
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1586
  >=65 years | 896
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.69 (11.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 626
  Male | 1856

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Incidence of the Composite Rate of Cardiac Death and Any Myocardial Infarction (MI) (Including Q-wave and Non-Q-wave)
Description: Cardiac death is defined as any death in which a cardiac cause cannot be excluded. (This includes but is not limited to acute myocardial infarction, cardiac perforation/pericardial tamponade, arrhythmia or conduction abnormality,cerebrovascular accident within 30 days of the procedure or cerebrovascular accident suspected of being related to the procedure, death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery).
  Myocardial Infarction (MI) - Q wave MI: Development of new, pathological Q wave on the ECG.
  -Non-Q wave MI: Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: 0 to 407 days
Population: Analysis Population exclude subjects who are truly lost-to-follow-up, defined as subjects who are lost to follow-up through given time point without any DMR event (all death, all MI, all revascularization) or stent thrombosis event.
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2391
Participants | 33

2. Primary Outcome: Number of Participants With Incidence of the Composite Rate of Cardiac Death and Any Myocardial Infarction (MI) (Including Q-wave and Non-Q-wave)
Description: as for outcome 1
Time Frame: 0 to 772 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2254
Participants | 55

3. Primary Outcome: Number of Participants With Incidence of the Composite Rate of Cardiac Death and Any Myocardial Infarction (MI) (Including Q-wave and Non-Q-wave)
Description: as for outcome 1
Time Frame: 0 to 1137 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2223
Participants | 63

4. Primary Outcome: Number of Participants With Incidence of the Composite Rate of Cardiac Death and Any Myocardial Infarction (MI) (Including Q-wave and Non-Q-wave)
Description: as for outcome 1
Time Frame: 0 to 1502 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2210
Participants | 76

5. Primary Outcome: Number of Participants With Incidence of the Composite Rate of Cardiac Death and Any Myocardial Infarction (MI) (Including Q-wave and Non-Q-wave)
Description: as for outcome 1
Time Frame: 0 to 1867 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2142
Participants | 84

6. Secondary Outcome: Number of Participants With Stent Thrombosis
Description: Definite Stent Thrombosis (ST) occurred by either angiographic/pathologic confirmation of ST.
  Angiographic confirmation:The presence of a thrombus that originates in the stent/in the segment 5mm proximal/distal to the stent&presence of at least 1 of the following criteria within 48hours:
  * Acute onset of ischemic symptoms at rest
  * New ischemic ECG changes
  * Typical rise&fall in cardiac biomarkers
  * Nonocclusive &occlusive thrombus
  Pathological confirmation:Evidence of recent thrombus within the stent determined at autopsy/via examination of tissue retrieved following thrombectomy.
  Probable ST may occur due to:
  * Unexplained death within first 30 days
  * Irrespective of the time after the index procedure,any MI that is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of ST&in the absence of any other obvious cause.
Time Frame: 0 to 1867 days
Population: Analysis Population exclude subjects who are truly lost-to-followup, defined as subjects who are lost to followup through given time point without any DMR event (all death, all MI, all revascularization) or stent thrombosis event.
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2142
Participants
  Definite | 5
  Definite & Probable | 10

7. Secondary Outcome: Number of Participants With Composite Rate of All Death, Any MI, and Any Repeat Revascularization
Description: All deaths includes
  * Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  * Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  * Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
  Myocardial Infarction (MI)
  * Q wave MI: Development of new, pathological Q wave on the ECG.
  * Non-Q wave MI: Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: 0 to 407 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2391
Participants | 90

8. Secondary Outcome: Number of Participants With Composite Rate of All Death, Any MI, and Any Repeat Revascularization
Description: as for outcome 7
Time Frame: 0 to 772 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2254
Participants | 154

9. Secondary Outcome: Number of Participants With Composite Rate of All Death, Any MI, and Any Repeat Revascularization
Description: as for outcome 7
Time Frame: 0 to 1137 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2223
Participants | 191

10. Secondary Outcome: Number of Participants With Composite Rate of All Death, Any MI, and Any Repeat Revascularization
Description: as for outcome 7
Time Frame: 0 to 1502 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2210
Participants | 235

11. Secondary Outcome: Number of Participants With Composite Rate of All Death, Any MI, and Any Repeat Revascularization
Description: as for outcome 7
Time Frame: 0 to 1867 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2142
Participants | 271

12. Secondary Outcome: Number of Participants With Composite Rate of Cardiac Death, MI Attributed to the Target Vessel (TV-MI), and All Target Lesion Revascularization (TLR)
Description: Cardiac Death:Cardiac death is defined as any death in which a cardiac cause cannot be excluded. (This includes but is not limited to acute myocardial infarction, cardiac perforation/pericardial tamponade, arrhythmia or conduction abnormality,cerebrovascular accident within 30 days of the procedure or cerebrovascular accident suspected of being related to the procedure, death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery).
  Target lesion revascularization is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion.
Time Frame: 0 to 407 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2391
Participants | 35

13. Secondary Outcome: Number of Participants With Composite Rate of Cardiac Death, MI Attributed to the Target Vessel (TV-MI), and All Target Lesion Revascularization (TLR)
Description: as for outcome 12
Time Frame: 0 to 772 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2254
Participants | 62

14. Secondary Outcome: Number of Participants With Composite Rate of Cardiac Death, MI Attributed to the Target Vessel (TV-MI), and All Target Lesion Revascularization (TLR)
Description: as for outcome 12
Time Frame: 0 to 1137 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2223
Participants | 71

15. Secondary Outcome: Number of Participants With Composite Rate of Cardiac Death, MI Attributed to the Target Vessel (TV-MI), and All Target Lesion Revascularization (TLR)
Description: as for outcome 12
Time Frame: 0 to 1502 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2210
Participants | 87

16. Secondary Outcome: Number of Participants With Composite Rate of Cardiac Death, MI Attributed to the Target Vessel (TV-MI), and All Target Lesion Revascularization (TLR)
Description: as for outcome 12
Time Frame: 0 to 1867 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2142
Participants | 95

17. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF) (Composite Rate of Cardiac Death, TV-MI and Ischemia-driven TLR)
Description: Target Lesion Failure is composite of Cardiac death/ Target Vessel Myocardial Infarction (TV-MI)/ Ischemic-Driven Target Lesion Revascularization (ID-TLR).
Time Frame: 0 to 407 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2391
Participants | 35

18. Secondary Outcome: Number of Participants With Target Lesion Failure (Composite Rate of Cardiac Death, TV-MI and Ischemia-driven TLR)
Description: as for outcome 17
Time Frame: 0 to 772 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2254
Participants | 60

19. Secondary Outcome: Number of Participants With Target Lesion Failure (Composite Rate of Cardiac Death, TV-MI and Ischemia-driven TLR)
Description: as for outcome 17
Time Frame: 0 to 1137 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2223
Participants | 69

20. Secondary Outcome: Number of Participants With Target Lesion Failure (Composite Rate of Cardiac Death, TV-MI and Ischemia-driven TLR)
Description: as for outcome 17
Time Frame: 0 to 1502 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2210
Participants | 85

21. Secondary Outcome: Number of Participants With Target Lesion Failure (Composite Rate of Cardiac Death, TV-MI and Ischemia-driven TLR)
Description: as for outcome 17
Time Frame: 0 to 1867 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2142
Participants | 93

22. Secondary Outcome: Number of Participants With Ischemia-driven Target Vessel Failure (ID-TVF) (Composite Rate of Cardiac Death, All MI and Target Vessel Revascularization (TVR))
Description: Ischemia-Driven Target Vessel Failure (TVF) is the composite endpoint comprised of
  * Cardiac death,
  * Myocardial infarction (Q wave and Non-Q wave),
  * Ischemia-driven target lesion revascularization by Coronary artery bypass grafting (CABG) or Percutaneous coronary intervention (PCI),
  * Ischemia-driven target vessel revascularization by CABG or PCI.
Time Frame: 0 to 407 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2391
Participants | 50

23. Secondary Outcome: Number of Participants With Ischemia-driven Target Vessel Failure (ID-TVF) (Composite Rate of Cardiac Death, All MI and Target Vessel Revascularization (TVR))
Description: as for outcome 22
Time Frame: 0 to 772 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2254
Participants | 86

24. Secondary Outcome: Number of Participants With Ischemia-driven Target Vessel Failure (ID-TVF) (Composite Rate of Cardiac Death, All MI and Target Vessel Revascularization (TVR))
Description: as for outcome 22
Time Frame: 0 to 1137 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2223
Participants | 100

25. Secondary Outcome: Number of Participants With Ischemia-driven Target Vessel Failure (ID-TVF) (Composite Rate of Cardiac Death, All MI and Target Vessel Revascularization (TVR))
Description: as for outcome 22
Time Frame: 0 to 1502 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2210
Participants | 123

26. Secondary Outcome: Number of Participants With Ischemia-driven Target Vessel Failure (ID-TVF) (Composite Rate of Cardiac Death, All MI and Target Vessel Revascularization (TVR))
Description: as for outcome 22
Time Frame: 0 to 1867 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2142
Participants | 136

27. Secondary Outcome: Number of Participants With Composite Rate of All Death and Any MI
Description: All deaths includes
  * Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  * Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  * Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
  Myocardial Infarction (MI)
  * Q wave MI Development of new, pathological Q wave on the ECG.
  * Non-Q wave MI Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: 0 to 407 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2391
Participants | 46

28. Secondary Outcome: Number of Participants With Composite Rate of All Death and Any MI
Description: as for outcome 27
Time Frame: 0 to 772 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2254
Participants | 80

29. Secondary Outcome: Number of Participants With Composite Rate of All Death and Any MI
Description: as for outcome 27
Time Frame: 0 to 1137 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2223
Participants | 92

30. Secondary Outcome: Number of Participants With Composite Rate of All Death and Any MI
Description: as for outcome 27
Time Frame: 0 to 1502 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2210
Participants | 120

31. Secondary Outcome: Number of Participants With Composite Rate of All Death and Any MI
Description: as for outcome 27
Time Frame: 0 to 1867 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2142
Participants | 137

32. Secondary Outcome: Number of Participants Experiencing Death
Description: Cardiac death is defined as any death in which a cardiac cause cannot be excluded. (This includes but is not limited to acute myocardial infarction, cardiac perforation/pericardial tamponade, arrhythmia or conduction abnormality,cerebrovascular accident within 30 days of the procedure or cerebrovascular accident suspected of being related to the procedure, death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery).
  - Non-cardiac death is defined as a death not due to cardiac causes (as defined above).
Time Frame: 0 to 407 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2391
Participants | 34

33. Secondary Outcome: Number of Participants Experiencing Death
Description: as for outcome 32
Time Frame: 0 to 772 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2254
Participants | 64

34. Secondary Outcome: Number of Participants Experiencing Death
Description: as for outcome 32
Time Frame: 0 to 1137 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2223
Participants | 75

35. Secondary Outcome: Number of Participants Experiencing Death
Description: as for outcome 32
Time Frame: 0 to 1502 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2210
Participants | 98

36. Secondary Outcome: Number of Participants Experiencing Death
Description: as for outcome 32
Time Frame: 0 to 1867 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2142
Participants | 113

37. Secondary Outcome: Number of Participants With Any MI
Description: Myocardial Infarction (MI):
  * Q wave MI: Development of new, pathological Q wave on the ECG.
  * Non-Q wave MI: Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: 0 to 407 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2391
Participants | 13

38. Secondary Outcome: Number of Participants With Any MI
Description: Myocardial Infarction (MI) - Q wave MI: Development of new, pathological Q wave on the ECG.
  -Non-Q wave MI: Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: 0 to 772 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2254
Participants | 20

39. Secondary Outcome: Number of Participants With Any MI
Description: as for outcome 38
Time Frame: 0 to 1137 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2223
Participants | 23

40. Secondary Outcome: Number of Participants With Any MI
Description: as for outcome 38
Time Frame: 0 to 1502 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2210
Participants | 28

41. Secondary Outcome: Number of Participants With Any MI
Description: as for outcome 38
Time Frame: 0 to 1867 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2142
Participants | 31

42. Secondary Outcome: Number of Participants With Revascularization
Description: Revascularization:
  * Target Lesion Revascularization (TLR) is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. The target lesion is defined as the treated segment from 5 mm proximal to the scaffold and to 5 mm distal to the test scaffold.
  * Target Vessel Revascularization (TVR) is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion.
  * Non Target Lesion Revascularization (Non-TLR) is any revascularization in the target vessel for a lesion other than the target lesion.
  * Non Target Vessel Revascularization (Non-TVR)is any revascularization in a vessel other than the target vessel.
Time Frame: 0 to 407 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2391
Participants | 49

43. Secondary Outcome: Number of Participants With Revascularization
Description: Revascularization:
  * Target Lesion Revascularization (TLR) is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. The target lesion is defined as the treated segment from 5 mm proximal to the scaffold and to 5 mm distal to the test scaffold.
  * Target Vessel Revascularization (TVR) is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion.
  * Non Target Vessel Revascularization (Non-TVR)is any revascularization in a vessel other than the target vessel.
Time Frame: 0 to 772 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2254
Participants | 83

44. Secondary Outcome: Number of Participants With Revascularization
Description: as for outcome 43
Time Frame: 0 to 1137 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2223
Participants | 111

45. Secondary Outcome: Number of Participants With Revascularization
Description: as for outcome 43
Time Frame: 0 to 1502 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2210
Participants | 132

46. Secondary Outcome: Number of Participants With Revascularization
Description: Revascularization:
  Target Lesion Revascularization (TLR) is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. The target lesion is defined as the treated segment from 5 mm proximal to the scaffold and to 5 mm distal to the test scaffold.
  Target Vessel Revascularization (TVR) is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion.
  Non Target Vessel Revascularization (Non-TVR)is any revascularization in a vessel other than the target vessel.
Time Frame: 0 to 1867 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2142
Participants | 154

47. Secondary Outcome: Number of Participants With Major Bleeding Complications (According to GUSTO Classification)
Description: Bleeding complications will be defined according to the GUSTO (Global Use of Strategies to Open Occluded Coronary Arteries) classification of severe, moderate, and mild bleeding events:
  * Severe or life-threatening: Either intracranial hemorrhage or bleeding that causes hemodynamic compromise and requires intervention.
  * Moderate: Bleeding that requires blood transfusion but does not result in hemodynamic compromise.
  * Mild: Bleeding that does not meet criteria for either moderate or severe bleeding.
Time Frame: 0 to 407 days
Population: Major Bleeding Complication analysed population excludes subjects who are truly lost-to-follow-up, defined as subjects who are lost to follow-up through given time point without any major bleeding complication event.
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2388
Participants | 14

48. Secondary Outcome: Number of Participants With Major Bleeding Complications (According to GUSTO Classification)
Description: Bleeding complications will be defined according to the GUSTO (Global Use of Strategies to Open Occluded Coronary Arteries) classification of severe, moderate, and mild bleeding events:
  Severe or life-threatening: Either intracranial hemorrhage or bleeding that causes hemodynamic compromise and requires intervention Moderate: Bleeding that requires blood transfusion but does not result in hemodynamic compromise Mild: Bleeding that does not meet criteria for either moderate or severe bleeding
Time Frame: 0 to 772 days
Population: as for outcome 47
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2231
Participants | 18

49. Secondary Outcome: Number of Participants With Major Bleeding Complications (According to GUSTO Classification)
Description: as for outcome 48
Time Frame: 0 to 1137 days
Population: as for outcome 47
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2160
Participants | 26

50. Secondary Outcome: Number of Participants With Major Bleeding Complications (According to GUSTO Classification)
Description: as for outcome 48
Time Frame: 0 to 1502 days
Population: as for outcome 47
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2126
Participants | 31

51. Secondary Outcome: Number of Participants With Major Bleeding Complications (According to GUSTO Classification)
Description: as for outcome 48
Time Frame: 0 to 1867 days
Population: as for outcome 47
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2029
Participants | 18

52. Secondary Outcome: Number of Participants Compliance With Dual Anti-platelet Therapy (DAPT)
Description: Dual Anti-platelet Therapy (DAPT) is Aspirin and Clopidogrel/Ticlopidine/Other.
Time Frame: 1 year
Population: Analysis population for each visit is the number of patients completed each protocol-required follow-up. Visit window± 42days.
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2384
Participants | 2231

53. Secondary Outcome: Number of Participants Compliance With Dual Anti-platelet Therapy (DAPT)
Description: Dual Anti-platelet Therapy (DAPT) is Aspirin and Clopidogrel/Ticlopidine/Other.
Time Frame: 2 years
Population: as for outcome 52
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2225
Participants | 1085

54. Secondary Outcome: Number of Participants Compliance With Dual Anti-platelet Therapy (DAPT)
Description: Dual Anti-platelet Therapy (DAPT) is Aspirin & Clopidogrel/Ticlopidine/Other.
Time Frame: 3 years
Population: as for outcome 52
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2151
Participants | 934

55. Secondary Outcome: Number of Participants Compliance With Dual Anti-platelet Therapy (DAPT)
Description: Dual Anti-platelet Therapy (DAPT) is Aspirin & Clopidogrel/Ticlopidine/Other.
Time Frame: 4 years
Population: as for outcome 52
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2116
Participants | 879

56. Secondary Outcome: Number of Participants Compliance With Dual Anti-platelet Therapy (DAPT)
Description: Dual Anti-platelet Therapy (DAPT) is Aspirin & Clopidogrel/Ticlopidine/Other.
Time Frame: 5 years
Population: as for outcome 52
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2029
Participants | 800

57. Secondary Outcome: Number of Participants With All Target Lesions Revascularization
Description: Target Lesion Revascularization (TLR) is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. The target lesion is defined as the treated segment from 5 mm proximal to the scaffold and to 5 mm distal to the test scaffold.
Time Frame: 0 to 407 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2391
Participants | 12

58. Secondary Outcome: Number of Participants With All Target Lesion Revascularization
Description: as for outcome 57
Time Frame: 0 to 772 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2254
Participants | 21

59. Secondary Outcome: Number of Participants With All Target Lesions Revascularization
Description: as for outcome 57
Time Frame: 0 to 1137 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2223
Participants | 25

60. Secondary Outcome: Number of Participants With All Target Lesion Revascularization
Description: as for outcome 57
Time Frame: 0 to 1502 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2210
Participants | 30

61. Secondary Outcome: Number of Participants With All Target Lesion Revascularization
Description: as for outcome 57
Time Frame: 0 to 1867 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2142
Participants | 33

62. Secondary Outcome: Number of Participants With All Target Vessel Revascularization
Description: Target Vessel Revascularization (TVR) is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion.
Time Frame: 0 to 407 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2391
Participants | 20

63. Secondary Outcome: Number of Participants With All Target Vessel Revascularization
Description: as for outcome 62
Time Frame: 0 to 772 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2254
Participants | 36

64. Secondary Outcome: Number of Participants With All Target Vessel Revascularization
Description: as for outcome 62
Time Frame: 0 to 1137 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2223
Participants | 42

65. Secondary Outcome: Number of Participants With All Target Vessel Revascularization
Description: as for outcome 62
Time Frame: 0 to 1502 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2210
Participants | 53

66. Secondary Outcome: Number of Participants With All Target Vessel Revascularization
Description: as for outcome 62
Time Frame: 0 to 1867 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 2142
Participants | 60

ADVERSE EVENTS:
Time Frame: 5 years
Description: Safety data was assessed based on the per protocol population (2482).
Arm/Group | Observational
All-Cause Mortality (participants affected / at risk) | 113/2482
Serious Adverse Events (participants affected / at risk) | 574/2482
Other Adverse Events (participants affected / at risk) | 113/2482
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Observational (N=2482)
Acute Heart Failure (Cardiac disorders) | 2
Acute Left Heart Failure (Cardiac disorders) | 1
Acute Left Ventricular Failure (Cardiac disorders) | 1
Acute Myocardial Infarction (AMI) (Cardiac disorders) | 4
Acute coronary syndrome (ACS) (Cardiac disorders) | 3
Acute coronary syndrome and heart failure (Cardiac disorders) | 1
Adams-Stokes Syndrome (Ventricular fibrillation (VF)) (Cardiac disorders) | 1
Angina (Cardiac disorders) | 121
Angina and Coronary Heart Disease (Cardiac disorders) | 3
Arrhythmia (Cardiac disorders) | 8
Atrial Fibrillation and Tachycardia (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrioventricular (AV) Block (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac Arrest (Cardiac disorders) | 3
Cardiac Function Insufficiency (Cardiac disorders) | 4
Cardiac Rupture (Cardiac disorders) | 1
Cardiac death (Cardiac disorders) | 2
Cardiogenic shock (Cardiac disorders) | 1
Cardiopulmonary disease (Cardiac disorders) | 1
Coronary Artery Disease recurrence (Cardiac disorders) | 5
Coronary Atherosclerotic Heart Disease (Cardiac disorders) | 3
Coronary Heart Disease (Cardiac disorders) | 56
Coronary artery disease (Cardiac disorders) | 8
Coronary artery revascularization (Cardiac disorders) | 2
Coronary heart disease worsened (Cardiac disorders) | 2
Heart Disease (Cardiac disorders) | 1
Heart Failure (Cardiac disorders) | 24
Ischemic cardiomyopathy (Cardiac disorders) | 1
Labor angina (Cardiac disorders) | 1
Left anterior descending (LAD) proximal stent occlusion (Cardiac disorders) | 1
Myocardial Infarction (Cardiac disorders) | 21
Non-ST segment elevation myocardial infarction (NSTEMI) (Cardiac disorders) | 6
Old Myocardial Infarction (Cardiac disorders) | 2
Palpitation (Cardiac disorders) | 7
Palpitation and Atrial fibrillation (Cardiac disorders) | 1
Paroxysmal Atrial Fibrillation (Cardiac disorders) | 2
Proximal right coronary artery (RCA) stenosis, not within the stent (Cardiac disorders) | 1
Sequelae of cerebral infarction (Cardiac disorders) | 1
Stable Angina (Cardiac disorders) | 11
Unstable Angina (Cardiac disorders) | 119
Ventricular Tachycardia (Cardiac disorders) | 1
Ventricular extrasystole (Cardiac disorders) | 1
Deaf (Ear and labyrinth disorders) | 1
Brain dysfunction (Endocrine disorders) | 1
Acute Gastroenteritis (Gastrointestinal disorders) | 2
Acute Intestinal Obstruction (Gastrointestinal disorders) | 1
Appendicitis (Gastrointestinal disorders) | 1
Biliary colic (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Gallstone (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
Gastrointestinal Bleeding (Gastrointestinal disorders) | 5
Incomplete intestinal obstruction (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Upper Gastrointestinal Bleeding (Gastrointestinal disorders) | 6
Abdominal Pain (General disorders) | 1
Atypical chest pain (General disorders) | 1
Bleeding Gums (General disorders) | 1
Chest Discomfort (General disorders) | 1
Chest Pain (General disorders) | 29
Chest Tightness (General disorders) | 25
Chest pain and chest tightness (General disorders) | 1
Colon Occupy (General disorders) | 1
Complex Ulcer Bleeding (General disorders) | 1
Death (General disorders) | 51
Hospitalization (General disorders) | 2
Hypovolemic Shock (General disorders) | 1
Intermittent Hemoptysis and Generalized Pain (General disorders) | 1
Intracranial Bleeding (General disorders) | 1
Low Back Pain (General disorders) | 1
Multiple Organ Failure (General disorders) | 4
Precordial discomfort (General disorders) | 1
Precordial pain (General disorders) | 1
Rehospitalization (General disorders) | 1
Severe bleeding complications (General disorders) | 1
Shortness of breath and Chest tightness (General disorders) | 1
Sick Sinus Syndrome (General disorders) | 2
Stomach bleeding (General disorders) | 7
Stent thrombosis (Vascular disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
GallStone And Cholecystitis (Hepatobiliary disorders) | 1
Common Cold (Infections and infestations) | 1
Otter disease (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2
Artery embolization (Injury, poisoning and procedural complications) | 1
Bone fracture (Injury, poisoning and procedural complications) | 1
Cerebral Hemorrhage (Injury, poisoning and procedural complications) | 12
Coronary artery revascularization and Coronary artery bypass grafting (Injury, poisoning and procedural complications) | 1
Distal Stent Restenosis (Injury, poisoning and procedural complications) | 1
Multiple rib fractures (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Non-Target Vessel Revascularization (Injury, poisoning and procedural complications) | 3
Percutaneous Coronary Intervention (PCI) (Injury, poisoning and procedural complications) | 2
Post-operative Percutaneous Coronary Intervention (PCI) (Injury, poisoning and procedural complications) | 5
Receiving catheter radiofrequency ablation (Injury, poisoning and procedural complications) | 1
Restenosis (Vascular disorders) | 5
Revascularization (Injury, poisoning and procedural complications) | 2
Stenosis (Vascular disorders) | 1
Stent Stenosis (Vascular disorders) | 1
Stent restenosis (Vascular disorders) | 2
Subarachnoid Hemorrhage (Injury, poisoning and procedural complications) | 2
Subdural Hematoma (Injury, poisoning and procedural complications) | 1
Upper Extremity Artery Stenosis (Vascular disorders) | 1
Diabetes (Metabolism and nutrition disorders) | 4
Newly Discovered Diabetes Mellitus (Metabolism and nutrition disorders) | 1
Type II Diabetes (Metabolism and nutrition disorders) | 3
Advanced Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Duodenal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Esophageal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intestinal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Kidney tumor metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Liver Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant Liver Tumors (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Right groin tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Stomach lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Throat Malignant Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral Infarction (Nervous system disorders) | 16
Cerebral Insufficiency (Nervous system disorders) | 1
Cerebral Thrombosis (Nervous system disorders) | 1
Convulsions (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Ischemic stroke (Nervous system disorders) | 1
Peripheral Neuropathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Acute pyelonephritis (Renal and urinary disorders) | 1
Kidney stones (Renal and urinary disorders) | 1
Prostate hyperplasia and urinary incontinence (Renal and urinary disorders) | 1
Renal Insufficiency (Renal and urinary disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2
Subcutaneous Bleeding (Skin and subcutaneous tissue disorders) | 1
All Coronary Revascularizations (Surgical and medical procedures) | 1
Coronary Artery Stenosis (Cardiac disorders) | 1
Coronary Stent Restenosis (Surgical and medical procedures) | 1
Heart surgery (Cardiac disorders) | 1
Hernia (General disorders) | 1
Blood pressure instability (Vascular disorders) | 1
Carotid Stenosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
Hypertension deterioration (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Observational (N=2482)
Abnormal liver enzymes (Hepatobiliary disorders) | 1
Angina (Cardiac disorders) | 11
Arrhythmia (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 2
Severe dizziness (Nervous system disorders) | 1
Bleeding (General disorders) | 5
Bleeding gums (General disorders) | 9
Blood in the stool (General disorders) | 2
Cardiac Troponin I (Ctni) Increased (Investigations) | 3
Cerebral Infarction (Nervous system disorders) | 1
Chest Pain (General disorders) | 6
Chest Tightness (General disorders) | 7
Chest Tightness and Chest Pain (General disorders) | 1
Congestive Heart Failure (Cardiac disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Diabetes (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Eye Bleeding (Eye disorders) | 1
Fundus Hemorrhage (Injury, poisoning and procedural complications) | 3
Gastric Ulcer (Gastrointestinal disorders) | 2
Gastrointestinal Bleeding (Gastrointestinal disorders) | 3
Gastrointestinal discomfort (Gastrointestinal disorders) | 1
Hand injury (Injury, poisoning and procedural complications) | 1
Heart Failure (Cardiac disorders) | 1
Hemoptysis (General disorders) | 1
Hemorrhoids (Injury, poisoning and procedural complications) | 1
Hypertension (Vascular disorders) | 1
Hyperthyroidism (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Increased myocardial enzymes (Investigations) | 2
Intermittent chest tightness (General disorders) | 1
Ischemic cardiomyopathy (Cardiac disorders) | 1
Labor angina (Cardiac disorders) | 2
Left Subconjunctival Hemorrhage (Injury, poisoning and procedural complications) | 1
Myocardial Infarction (Cardiac disorders) | 1
Myocardial hypertrophy (Cardiac disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Nose bleeding (General disorders) | 2
Occult blood (General disorders) | 1
Ocular hyperemia (Eye disorders) | 1
Positive occult blood test (Investigations) | 1
Postoperative Cardiac Troponin I (Ctni) Increased (Investigations) | 1
Postoperative Troponin I (TnI) Increased (Investigations) | 3
Right Femoral Vein Thrombosis (Vascular disorders) | 1
Right lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Severe palpitation (Cardiac disorders) | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2
Side effects of Aspirin (Injury, poisoning and procedural complications) | 1
Sinus Bradycardia (Cardiac disorders) | 1
Skin Bruises (Skin and subcutaneous tissue disorders) | 3
Skin ecchymosis (Skin and subcutaneous tissue disorders) | 1
Stable angina (Cardiac disorders) | 3
Stomach Bleeding (Gastrointestinal disorders) | 4
Stomach discomfort (General disorders) | 1
Stomach pain (General disorders) | 2
Subcutaneous Bleeding (Injury, poisoning and procedural complications) | 1
Throat bleeding (General disorders) | 1
Unstable Angina (Cardiac disorders) | 4
Upper Gastrointestinal Bleeding (Gastrointestinal disorders) | 2
Upper abdominal discomfort (Gastrointestinal disorders) | 1
Upper gastrointestinal bleeding (Gastrointestinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less